CLINICAL TRIAL: NCT02406755
Title: H-SENSES PROJECT Self Care Mediated by the Senses: Assessing the Impact on Self-esteem, Stress and Well-being of Female Health Professionals
Brief Title: H-Senses Project - Self Care Mediated by the Senses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Eliseth Ribeiro Leao, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-Senses
Record Dates: First submitted 2014-10-27; First posted 2015-04-02 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): This control group will not receive an intervention.
- one-sensory self care (Active Comparator): Daily moisturizing body care with an odorless moisturizer (Todo Dia® - Natura) for 30 days.
  Interventions: Other: one-sensory self care (Todo Dia®)
- bi-sensory self care (Active Comparator): Daily moisturizing body care with a moisturizer with cotton fragance (Todo Dia® - Natura) for 30 days.
  Interventions: Other: bi-sensory self care (Todo Dia®)
- multisensory self care (Active Comparator): Daily moisturizing body care with a moisturizer with cotton fragance (Todo Dia® - Natura) for 30 days, and will watch a video with music and images of nature during self-care.
  Interventions: Other: multisensory self care (Todo Dia®)

INTERVENTIONS:
Other: one-sensory self care (Todo Dia®) — daily use of odorless body moisturizer (Todo Dia® - Natura)
  Arms: one-sensory self care
Other: multisensory self care (Todo Dia®) — daily use of moisturizing body with cotton fragrance (Todo Dia® - Natura) + audiovisual stimulus
  Arms: multisensory self care
Other: bi-sensory self care (Todo Dia®) — daily use of moisturizing body with cotton fragrance (Todo Dia® - Natura)
  Arms: bi-sensory self care

SUMMARY:
Randomized clinical trial about self-care mediated by the senses in female health professionals and their influence on stress, self-esteem, mood states, life satisfaction and levels of salivary cortisol.

DETAILED DESCRIPTION:
The work environment of health professionals is commonly considered stressful, given that they need to deal with difficult situations that include pain, risk of death, the decisions that need to be fast and accurate, and conflicts generated in interpersonal relationships. There is an ongoing discussion that the investigators need to care for those who care, however, there are few interventions studied and validated to effectively reduce the stress of these professionals that resonate in states of well-being. There is little room for discussion of this topic during the workday, as well as to learn techniques and measures for effective stress management. This study aims to explore the relationship between well-being, self-esteem and stress of women health professionals, and compare three self-care interventions mediated by the senses.

ELIGIBILITY:
Inclusion Criteria:

* Professional healthcare;
* working in healthcare or administrative area in hospital
* Voluntary participation;
* Signed in term of free and informed consent.

Exclusion Criteria:

* Evaluation with relevant dermatological findings diagnosed by a dermatologist;
* Work at nighttime or in alternate periods (because of known chronobiological changes that would affect the study of cortisol, one of the outcomes considered in the study);
* who are breastfeeding;
* Be pregnant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress (Lipp Stress Inventory and Symptoms of Stress List) | baseline, 30 days, 60 days
  Lipp Stress Inventory and Symptoms of Stress List

SECONDARY OUTCOMES:
Change in cortisol levels | baseline, 30 days, 60 days
  Saliva will be collected to measure cortisol levels: 7-9 am

OTHER OUTCOMES:
Changes in Satisfaction with life (Satisfaction With Life Scale) | baseline, 30 days, 60 days
  Satisfaction With Life Scale
Changes in Positive and Negative Affective | baseline, 30 days, 60 days
  Positive and negative affect scale
Change in perceived self-esteem (Rosenberg's self-esteem Scale) | baseline, 30 days, 60 days
  Rosenberg's self-esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein - Albert Einstein Jewish Institute for Education and Research
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ribeiro VF, Filho CF, Valenti VE, Ferreira M, de Abreu LC, de Carvalho TD, Xavier V, de Oliveira Filho J, Gregory P, Leao ER, Francisco NG, Ferreira C. Prevalence of burnout syndrome in clinical nurses at a hospital of excellence. Int Arch Med. 2014 May 9;7:22. doi: 10.1186/1755-7682-7-22. eCollection 2014. PMID 24860618
- [Background] Caminha LB, da Silva MJ, Leao ER. [The influence of musical rhythms on the perception of subjective states of adult patients on dialysis]. Rev Esc Enferm USP. 2009 Dec;43(4):923-9. doi: 10.1590/s0080-62342009000400026. Portuguese. PMID 20085165
- [Derived] Leao ER, Dal Fabbro DR, Oliveira RB, Santos IR, Victor ED, Aquarone RL, Andrade CB, Ribeiro VF, Oliveira RC, Friedlander R, Ferreira DS. Stress, self-esteem and well-being among female health professionals: A randomized clinical trial on the impact of a self-care intervention mediated by the senses. PLoS One. 2017 Feb 27;12(2):e0172455. doi: 10.1371/journal.pone.0172455. eCollection 2017. PMID 28241070